CLINICAL TRIAL: NCT00509158
Title: Phase I and IIa Trial for Assessment of Safety, Immunogenicity and Efficacy Against Sporozoite Challenge of the Candidate Malaria Vaccine PfLSA-3-rec
Brief Title: Safety and Efficacy Study of Plasmodium Falciparum LSA-3 Malaria Vaccine
Acronym: LSA-3-rec
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Institut Pasteur (Industry)
Responsible Party: Prof. dr. R.W. Sauerwein, principle investigator, Radboud University Nijmegen Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LSA3_01_06
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Last update posted 2010-02-23 (Estimated); Status verified 2008-11

CONDITIONS: Healthy
Keywords: safety; immunogenicity; efficacy
MeSH Terms: interventions — Aluminum Hydroxide; Adjuvants, Pharmaceutic; mannide monooleate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: arm I: PfLSA-3-rec with aluminium hydroxide as adjuvant
Biological: arm 2: PfLSA-3-rec with Montanide Isa 720 as adjuvant

SUMMARY:
Malaria is responsible for over 2 million deaths each year. The development of an efficient vaccine would present by far the best solution for solving this disastrous situation. Liver-Stage-Antigen-3 (LSA-3) is an antigen that is mainly exhibited by Plasmodium falciparum sporozoites and liver-stage parasites. It is characterized by its remarkable antigenicity in humans with a wide range and a variety of B and T-lymphocyte epitopes, by its extremely high immunogenicity and by an excellent protective efficacy against sporozoite challenge in animal models. Therefore, PfLSA-3-rec is a promising candidate vaccine against P. falciparum in humans The aim is to screen two different formulations of the recombinant malaria vaccine PfLSA-3-rec, one adjuvated with aluminium hydroxide and one with Montanide Isa 720, by assessing the safety and immunogenicity (phase I) profile of each formulation in humans, as well as its protective efficacy following a sporozoite challenge (phase IIa).

ELIGIBILITY:
(Main) Inclusion Criteria:

* Male and female age ≥18 and ≤ 45 years
* Good general health based on history, physical en laboratory examination
* Available for and willingness to undergo a P. falciparum sporozoite challenge following the immunization course
* Resident near the Radboud University Medical Center Nijmegen, having 24h access to a telephone
* Living with a third party that could contact the clinicians in case of alteration of conscience
* Agreement to refrain from blood donation during the course of the study and afterwards
* Negative pregnancy test and the use of effective contraception during the whole study period

(Main) Exclusion Criteria:

* Any history of malaria
* Known exposure to malaria in the previous 6 months, defined as a visit to a malaria-endemic region.
* Planned to travel to endemic malaria areas during the study period
* Prior administration of an investigational malaria vaccine
* Administration of a vaccine or gammaglobulin not foreseen by the clinical trial protocol within 30 days prior to the first immunization and up to six months after the last immunization.
* Participation in any other clinical trial within 90 days prior to the onset of the trial or more than four clinical trials in the past year
* The use of chronic immunosuppressive drugs or other immune modifying drugs within three months of vaccination (inhaled and topical corticosteroids are allowed)
* Positive serological tests for P falciparum (LSA-3) ELISA and/or a positive P. falciparum PCR
* Known hypersensitivity to vaccine components
* Contra-indications to Riamet® including treatment taken by the volunteers that interfere with Riamet® (e.g. concurrent use of medicines that prolong QT-interval)
* Symptoms, physical signs and laboratory values suggestive of systemic disorders, including renal, hepatic, cardiovascular, pulmonary, skin, immunodeficiency, psychiatric and other conditions, which could interfere with the interpretation of the study results or compromise the health of the volunteers
* An estimated, ten year risk of fatal cardiovascular disease of ≥5%, as estimated by the Systematic Coronary Risk Evaluation (SCORE) system.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Phase I: proportion and severity of adverse events in both intervention groups. | 1 year from first immunization
Phase IIa: proportion of volunteers reaching day 21 post-infection without or with a delayed onset of parasitemiae compared to control group (parasetimiae defined as ≥2 parasites per 200 fields in a thick blood film). | 6 weeks from sporozoite challenge

SECONDARY OUTCOMES:
Phase I and IIa: Immunogenicity evaluation: antibody and cellular responses to vaccination with PfLSA-3-rec vaccine formulations. | 1 year from first immunization
Phase IIa: The length of time (in hours) between parasite inoculation and detection of parasitemia, if any, up to 21 days. | 6 weeks from sporozoite challenge

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sauerwein, Prof MD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Derived] Coffeng LE, Hermsen CC, Sauerwein RW, de Vlas SJ. The Power of Malaria Vaccine Trials Using Controlled Human Malaria Infection. PLoS Comput Biol. 2017 Jan 12;13(1):e1005255. doi: 10.1371/journal.pcbi.1005255. eCollection 2017 Jan. PMID 28081133